CLINICAL TRIAL: NCT00201058
Title: Tailored Asthma Management for Urban Teens
Acronym: Puff City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christine Joseph, Senior Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1299; R01HL068971-04 (NIH); R01HL068971 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: urban; adolescents; African American; web-based; computer tailoring; school based
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Receives tailored web-based program
  Interventions: Behavioral: Tailored Web-based Asthma Management
- 2 (Active Comparator): Control students receive existing web-based, generic asthma education
  Interventions: Behavioral: Generic web-based asthma education

INTERVENTIONS:
Behavioral: Tailored Web-based Asthma Management — Web-based asthma management
  Arms: 1
Behavioral: Generic web-based asthma education — 4 computer sessions over a period of 180 days
  Arms: 2

SUMMARY:
The purpose of this project is to refine and further evaluate an online asthma management and education program for urban teenagers. This project is a continuation of Puff City I, a project piloting and evaluating a tailored, school-based, computerized asthma education program for urban teenagers. In this second phase of research, a new version of software (Puff City II) will be created that will target resistance to change and relapse, and using a tested, theory-based approach to student recruitment, conduct a randomized trial to test the efficacy of this new software.

DETAILED DESCRIPTION:
BACKGROUND:

Teenagers are among an age group that has seen dramatic increases in deaths from asthma. In Detroit, asthma death rates for teenagers are high relative to younger ages, despite a higher prevalence in the latter age group. Early studies suggest that inadequate asthma management plays a significant role in these grim statistics.

DESIGN NARRATIVE:

The study hypothesis is that students randomized to the intervention group will have lower asthma-related morbidity as determined by fewer emergency department visits and hospitalizations at the time of the 12-month follow-up. Based on a second hypothesis of better functional status among students randomized to the intervention group, secondary outcomes include fewer symptom-days, symptom-nights, school days missed, and days of restricted activity at the time of the 12-month follow-up. In addition, it is hypothesized that students in the intervention group will have higher scores on the Juniper Pediatric Quality of Life scale at 12 months. Finally, it is hypothesized that intervention students would exhibit positive changes in adherence behavior, having a rescue inhaler nearby, and smoking at the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosis of asthma AND recent asthma symptoms, health care utilization for asthma, and/or use of medication (or refills of medication) to alleviate asthma symptoms OR
* No physician diagnosis of asthma AND positive responses to items selected from the International Study of Asthma and Allergy in Children (ISAAC) survey AND asthma symptoms similar to those used in the Expert Panel II for classification of mild intermittent asthma

Exclusion Criteria:

* Does not meet asthma symptom criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Asthma-related morbidity | Measured at baseline, 6 months, and 12 months with the latter being the timepoint of interest

SECONDARY OUTCOMES:
Symptom-days | Measured at baseline, 6 months, and 12 months with the latter being the timepoint of interest
Symptom-nights | Measured at baseline, 6 months, and 12 months with the latter being the timepoint of interest
School days missed | Measured at baseline, 6 months, and 12 months with the latter being the timepoint of interest
Days of restricted activity | Measured at baseline, 6 months, and 12 months with the latter being the timepoint of interest

CONTACTS AND LOCATIONS:
Overall Officials: Christine Joseph, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Joseph CL, Havstad S, Johnson CC, Vinuya R, Ownby DR. Agreement between teenager and caregiver responses to questions about teenager's asthma. J Asthma. 2006 Mar;43(2):119-24. doi: 10.1080/02770900500498246. PMID 16517427
- [Background] Joseph CL, Havstad S, Anderson EW, Brown R, Johnson CC, Clark NM. Effect of asthma intervention on children with undiagnosed asthma. J Pediatr. 2005 Jan;146(1):96-104. doi: 10.1016/j.jpeds.2004.09.001. PMID 15644831
- [Background] Joseph CL, Williams LK, Ownby DR, Saltzgaber J, Johnson CC. Applying epidemiologic concepts of primary, secondary, and tertiary prevention to the elimination of racial disparities in asthma. J Allergy Clin Immunol. 2006 Feb;117(2):233-40; quiz 241-2. doi: 10.1016/j.jaci.2005.11.004. PMID 16461121
- [Result] Joseph CL, Baptist AP, Stringer S, Havstad S, Ownby DR, Johnson CC, Williams LK, Peterson EL. Identifying students with self-report of asthma and respiratory symptoms in an urban, high school setting. J Urban Health. 2007 Jan;84(1):60-9. doi: 10.1007/s11524-006-9121-y. PMID 17200800
- [Result] Joseph CL, Peterson E, Havstad S, Johnson CC, Hoerauf S, Stringer S, Gibson-Scipio W, Ownby DR, Elston-Lafata J, Pallonen U, Strecher V; Asthma in Adolescents Research Team. A web-based, tailored asthma management program for urban African-American high school students. Am J Respir Crit Care Med. 2007 May 1;175(9):888-95. doi: 10.1164/rccm.200608-1244OC. Epub 2007 Feb 8. PMID 17290041
- [Result] Joseph CL, Havstad SL, Ownby DR, Zoratti E, Peterson EL, Stringer S, Johnson CC. Gender differences in the association of overweight and asthma morbidity among urban adolescents with asthma. Pediatr Allergy Immunol. 2009 Jun;20(4):362-9. doi: 10.1111/j.1399-3038.2008.00803.x. Epub 2008 Sep 22. PMID 18823359
- [Derived] Ezell JM, Saltzgaber J, Peterson E, Joseph CL. Reconnecting with urban youth enrolled in a randomized controlled trial and overdue for a 12-month follow-up survey. Clin Trials. 2013 Oct;10(5):775-82. doi: 10.1177/1740774513498320. Epub 2013 Aug 27. PMID 23983157
- [Derived] Joseph CL, Ownby DR, Havstad SL, Saltzgaber J, Considine S, Johnson D, Peterson E, Alexander G, Lu M, Gibson-Scipio W, Johnson CC; Research team members. Evaluation of a web-based asthma management intervention program for urban teenagers: reaching the hard to reach. J Adolesc Health. 2013 Apr;52(4):419-26. doi: 10.1016/j.jadohealth.2012.07.009. Epub 2012 Sep 27. PMID 23299008
- [Derived] Guglani L, Havstad SL, Johnson CC, Ownby DR, Joseph CL. Effect of depressive symptoms on asthma intervention in urban teens. Ann Allergy Asthma Immunol. 2012 Oct;109(4):237-242.e2. doi: 10.1016/j.anai.2012.07.010. Epub 2012 Aug 15. PMID 23010228
- [Derived] Joseph CL, Saltzgaber J, Havstad SL, Johnson CC, Johnson D, Peterson EL, Alexander G, Couper MP, Ownby DR. Comparison of early-, late-, and non-participants in a school-based asthma management program for urban high school students. Trials. 2011 Jun 6;12:141. doi: 10.1186/1745-6215-12-141. PMID 21645394